CLINICAL TRIAL: NCT03100487
Title: Efficacy of Remote Audio Recorded Guided Imagery vs Deep Breathing Exercises on Primary Pediatric Care Patients With Functional Gastrointestinal Pain Disorders (TCH Pediatric Pilot Award)
Brief Title: Efficacy of Audio Recorded Guided Imagery vs Deep Breathing Exercises on Functional Gastrointestinal Pain Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, John Hollier, Assistant Professor, Pediatrics-Gastroenterology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-39390
Record Dates: First submitted 2017-01-19; First posted 2017-04-04 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Abdominal Pain; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Abdominal Pain; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Audio Record Guided Imagery (ARGI) (Experimental): The audio recorded guided imagery sessions (treatment) will be delivered through a digital audio player (Apple iPod Shuffle).
  Interventions: Device: Apple iPod Shuffle
- Deep Breathing Exercises (Experimental): The deep breathing exercises (control) will be delivered through a digital audio player (Apple iPod Shuffle).
  Interventions: Device: Apple iPod Shuffle

INTERVENTIONS:
Device: Apple iPod Shuffle — One session at least 5 days a week for a total of 8 weeks

SUMMARY:
The purpose of this study is to:

1. Determine if audio recorded guided imagery vs deep breathing exercises delivered via a digital media player improves abdominal pain symptoms in children with functional gastrointestinal pain disorders managed in the primary care setting.
2. Determine if audio recorded guided imagery and deep breathing exercises delivered via a digital media player improves psychosocial distress in children affected by functional gastrointestinal pain disorders managed in the primary care setting.

The possibility of treating functional gastrointestinal pain disorders using remotely delivered psychosocial therapies has the potential to treat many children affected by functional gastrointestinal pain disorders in a cost-effective manner. This study will provide insight into how well these patients in the primary care could benefit from such interventions.

DETAILED DESCRIPTION:
Children managed in primary care with a functional gastrointestinal pain disorder will be recruited and studied for this trial. After participants are deemed eligible, they will complete multiple questionnaires and then be randomly assigned (like a flip of a coin) to either guided imagery or deep breathing exercises delivered via a digital media player. Participants will be instructed to listen to the tracks at least 5 days per week for an 8 week intervention period.

At week 3 of the intervention period, the participant will complete another 2 week pain and stool diary.

At week 7 of the intervention period, the participant will complete another 2 week pain and stool dairy. After this diary is completed, the participant will again complete multiple questionnaires for their final visit.

ELIGIBILITY:
Inclusion Criteria:

1. Children who meet criteria for a functional gastrointestinal pain disorder.
2. Children who manage their abdominal pain in the primary care setting.

Exclusion Criteria:

1. Children who have other comorbidities that are associated with chronic abdominal pain including abdominal surgery and other medical diagnoses that can cause chronic abdominal pain.
2. Children with an intellectual disability which would hamper their ability to communicate with study staff about their pain and complete study questionnaires.
3. Children who have presented to a gastroenterologist for abdominal pain management
4. Children who have previously used deep breathing exercises or guided imagery to manage their abdominal pain.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change in abdominal pain symptoms | Change from Baseline to 8 weeks post-treatment
  Abdominal Pain Index

SECONDARY OUTCOMES:
Improvement in health-related quality of life | Change from Baseline to 8 weeks post-treatment
  Pediatric Quality of Life Inventory (Peds QL) Questionnaire
Change in Psychosocial Distress | Change from Baseline to 8 weeks post-treatment
  Behavior Assessment System for Children (BASC 3) Questionnaire
Adherence to Intervention | 8 weeks after treatment
  Count of Number of Sessions Played

CONTACTS AND LOCATIONS:
Overall Officials: John M Hollier, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No